CLINICAL TRIAL: NCT02033499
Title: Effect of Glucose Monitoring on Patient and Provider Outcomes in Non-insulin Treated Diabetes
Brief Title: Three Approaches to Glucose Monitoring in Non-insulin Treated Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Katrina Donahue, MD, MPH, Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2047
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-05

CONDITIONS: DIABETES MELLITUS, NONINSULIN-DEPENDENT, 2 (Disorder)
Keywords: Blood Glucose Self-Monitoring; Self-Monitoring, Blood Glucose; Diabetes Mellitus, Type 2; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigators including the bio-statistician were blind to the study assignment.
Oversight: Data Monitoring Committee: No

ARMS (3):
- No testing (No Intervention): No testing
- standard messaging (Other): SMBG standard messaging
  Interventions: Behavioral: SMBG
- enhanced messaging (Other): SMBG enhanced messaging
  Interventions: Behavioral: SMBG

INTERVENTIONS:
Behavioral: SMBG — Blood glucose levels are tested once daily.
  Other Names: Self-monitoring of blood glucose with a Telcare glucometer
  Arms: enhanced messaging; standard messaging

SUMMARY:
For the nearly 75% of patients living with type 2 diabetes (T2DM) that do not use insulin, decisions regarding self-monitoring of blood glucose (SMBG) are unclear. SMBG testing is a resource intensive activity without firmly established patient benefits. While SMBG holds great promise for sparking favorable behavior change, the potential for no benefit or even patient harm must be acknowledged. Possible negative effects on patient quality of life must be more closely examined along with the speculative benefits of SMBG in non-insulin treated T2DM. Among studies examining this issue a general consensus is evolving; while SMBG may or may not be useful, its value can only be fully appreciated when the SMBG results are provided to patients in a useful manner. The overarching goal of this proposal is to assess the impact of three different SMBG testing approaches on patient-centered outcomes in patients with non-insulin treated T2DM within the real-world, clinic setting. In this pragmatic trial, 450 patients will be randomized to one of the following three SMBG testing regimens: 1) no SMBG testing, 2) once daily SMBG testing with standard patient feedback consisting of glucose values being immediately reported to the patient through the glucose meter, and 3) once daily SMBG testing with enhanced patient feedback consisting of glucose values being immediately reported to the patient plus automated, tailored feedback messaging. The first two arms represent common SMBG testing approaches. The third arm is an enhanced, patient-centered approach to SMBG testing. SMBG values will be evaluated at routine clinic visits over 52 weeks.

DETAILED DESCRIPTION:
Within the context of a controlled and randomized but pragmatic trial, we seek to answer the following question: does SMBG testing make sense for Non-insulin treated (NIT) diabetes mellitus (DM) patients in terms of either A1c values or Health-related Quality of Life (QOL). We will also examine whether or not patients with different baseline characteristics might see different outcomes from three SMBG testing approaches. To achieve our goal of testing SMBG options in community-based primary care practices, the study has been designed to minimize as much as possible any interruptions in or alterations to standard daily patient care. We will recruit 450 patients from five primary care practices. Patients will be followed for one year. During routine clinic visits, their health care providers will be guided to modify therapies based on American Diabetes Association (ADA) guidelines, which focus on A1c values and SMBG values if available.

Study Arms Two of the three study arms were chosen to reflect existing, widely used options for patients with NIT DM. Arm 3, described below, of this trial is particularly novel in that it tests the potential benefit of new technology now available to these patients; namely, wireless transmission of blood glucose test results accompanied by instantaneous tailored feedback. While this option may hold great promise for patients and their providers, data supporting this are lacking. The results of this study will inform consumers and providers about whether this new technology can support efforts to alter behaviors in a way that results in improved A1c values or better quality of life. Particularly appealing is that this approach employs technology that supports more efficient use of SMBG values by both patients and their providers. In terms of their pragmatic 'fit', all three groups fit easily into current practice at the participating practices. For example, they do not require extra clinic visits (other than possibly the initial recruitment assessment), and while staff will need to download glucose reports for patients in Arms 2 and 3, this will be a very simple, streamlined procedure. In terms of risks to patients, none of the three groups puts patients at any additional risk, because all three are versions of 'standard practice' for this patient population and doctors are free to alter therapies and testing schedules as they normally would.

* Arm 1: No SMBG Testing This group represents an approach to SMBG that is supported by research and followed by many primary care providers. Patients randomized to this group will not be provided a meter, but will receive standardized education detailing the signs and symptoms of hyper- and hypoglycemia and information regarding lifestyle approaches for the maintenance of normoglycemia. If they have previously been obtaining SMBG values, they will be asked to discontinue. Healthcare providers and staff will be alerted that these patients are in the no testing arm and will be encouraged to maintain treatment fidelity except where patient safety is a concern. Study coordinators will provide patients with both written and oral educational information supporting the approach of no SMBG testing, with a view toward reconciling any messages they may have received in the past or will receive in the future regarding SMBG. This education will recur every 3-6 months at routine clinic visits (the recommended follow-up frequency for persons with T2DM) by their health care providers. A1c will be obtained during these visits as per usual care and providers will adjust medication and lifestyle recommendations as they see fit. Providers will be given an algorithm based on current ADA recommendations relating to A1c results to use as a guide for treatment modification.
* Arm 2: Once Daily Testing with Standard Feedback This group represents an approach taken by a large proportion of NIT DM patients in the US. At the assessment visit, patients will be given the study glucose meter and testing supplies, along with instruction for their use. They will be asked to test once daily and at different times of the day on a rotating basis, in order to obtain a representative distribution of blood glucose values over time. The meter will have wireless capability such that it will transmit both the SMBG result and the time of testing to a secure server. Subjects will also note the circumstances of their test times on the glucose meter (e.g., fasting, 2 hours post meal, etc.) and this information will also be sent to the server. As with Arm 1, Arm 2 patients will receive training in hyper- and hypoglycemia and approaches for maintaining normoglycemia. They will also receive training and written material instructing them in how to interpret their SMBG readings and actions they might take in response to those values. SMBG results will be reviewed at all clinic visits (3-6 month intervals) by the primary care provider using a print out of glucose meter values downloaded and analyzed wirelessly. During the early phase of the project, a streamlined system will be developed to allow participating clinic staff to download the SMBG values with minimal effort and create the accompanying SMBG report for the patient's provider. This customized report, detailing blood glucose averages, ranges and standard deviations, will be generated for all group 2 participants and given to their provider prior to each routine clinic visit. The report will identify problematic glucose values (hypo- and hyperglycemia) and suggested approaches for addressing these problems. Providers will review the results with the participant and make appropriate treatment recommendations based upon blood glucose trends. The recommendations in the report will be driven by an algorithm for treatment modification based upon ADA guidelines which will include suggestions for both lifestyle and pharmacotherapy adjustments. At the end of each clinic visit, patients will be instructed by their primary care provider to continue once daily testing. Using shared decision-making and standardized testing recommendations, the health care provider and the patient will jointly determine the testing approach (e.g., timing of once daily testing) the patient will employ over the next monitoring period.
* Arm 3: Once Daily Testing with Enhanced Feedback This Arm represents an enhanced, patient-centered approach. Participants randomized to Arm 3 will, like the Arm 2 participants, be instructed to test once daily and at different times of the day, and their glucose values will be transmitted wirelessly to a server. However, for Arm 3 participants, the blood glucose values will be analyzed automatically each time a value is transmitted. Based upon the value, instantaneous personalized feedback will be provided via wireless messaging to the patients' glucose meters. These messages will not include suggestions for pharmacological therapy modification but will be motivational in nature, including suggestions to enhance efforts at lifestyle management and adherence to pharmacologic therapy if prescribed. At weekly intervals, an analysis of the SMBG values from the previous week will be sent to the glucose meter highlighting trends and identifying specific problematic times. Subjects will also receive messages reminding them of upcoming clinic visits (beginning 1 week prior to their scheduled visit). As with Arm 2, SMBG results and customized reports will be downloaded and reviewed at all clinic visits by the primary care provider. In addition, a summary of the messages sent wirelessly to the patient since the most recent visit will be included. Like the glucose values report, this message report will be given to all providers at the beginning of the clinic visit and providers will be asked to also review these results with the patient. Providers will make appropriate treatment recommendations based upon blood glucose trends and messages. Report recommendations will be driven by an algorithm for treatment modification based upon ADA treatment guidelines and include suggestions for lifestyle and pharmacotherapy adjustments. At the end of the clinic visit, patients will be instructed by their primary care provider to continue testing their blood glucose once daily and collaboratively determine the testing approach (e.g., timing of once daily testing) the patient will employ over the next monitoring period.

Potential Alterations to the Testing Recommendations: Providers will be strongly encouraged to maintain SMBG testing fidelity based upon the treatment arm to which a patient is randomized; however, if a provider believes that testing should occur more frequently due to concern for serious unrecognized hypo- or hyperglycemia or for any other reason, testing recommendations may be modified. This approach provides for patient safety and preserves the pragmatic nature of the trial. Glucose testing strips will be provided to participants on a quarterly basis. If a provider deems that SMBG testing should occur more frequently than what is recommended to the patient based on the study arm to which he or she has been randomized, the health care provider must write the prescription for the additional test strips and the strips must be paid for out-of-pocket or through insurance. Following an intention to treat model, patients who opt not to follow the testing regimen to which they were randomly assigned will be encouraged to remain in the study. Any deviations from the assigned SMBG testing protocol will be readily known via the glucose meter reports.

Mixed methods approach. A mixed methods approach in which both qualitative and quantitative data are collected provides advantages when exploring complex research questions such as the ones posed in this proposal. The quantitative data will allow us to assess changes in objective measures, while the qualitative data will provide a deeper understanding of patients' and providers' experiences with the various components of SMBG testing arms (e.g., the meters, SMBG results, personalized messaging, downloadable reports, treatment algorithms, etc.) It is also the case that, while some patients are interested in seeing hard facts and figures, others prefer testimonials from patients like themselves. The mixed methods approach enables us to provide both types of information, increasing the effectiveness and uptake of our dissemination efforts.

Recruitment and randomization procedures. Patient Recruitment: All potentially eligible patients expressing interest in the study will complete an initial screening phone call. The call will take about 15 minutes, during which a member of the study team will describe the study, answer questions, and conduct a short set of simple screening to determine eligibility. Eligible patients who remain interested in participation will complete an assessment visit with a research coordinator. To decrease patient burden and further engage participating practices, assessment visits will occur at the patient's primary care office. Assessments will be separate from their appointment with their primary care provider, and may or may not occur on the same day as a regularly scheduled clinic visit, though for patient convenience we will make every effort to coordinate the assessments with a regular clinic visits. During these assessments, the research coordinator will review the study details in greater depth, verify all inclusion and exclusion criteria, and obtain written informed consent.

Patient Randomization: After providing informed consent, baseline A1c, and completing all baseline study questionnaires, participants will be randomized to one of the three arms using sequentially numbered, opaque, sealed envelopes. The research coordinator will review the treatment assignment with the patient, using a standardized script, provide the training and supplies necessary for participation in that study arm and answer any remaining questions.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 2 diabetes
* Age > 30
* An established patient at the participating UNC Physicians Network (UNCPN) practice who identifies a UNCPN health care provider within that practice as their primary provider of diabetes care.
* A1c >6.5% but <9.5% within the 6 months preceding the screening call/visit, as obtained from the patient's medical record.
* Willing to comply with the results of random assignment into a study group.

Exclusion Criteria:

* Currently sees or plans to see an endocrinologist or other diabetes specialist in the next year.
* Use of insulin
* Is or plans to become pregnant in the next 12 months.
* Plans to relocate in the next 12 months.
* Has other conditions (e.g. renal or cardiovascular disease, poor visual acuity), other factors (e.g. frailty,) or comorbidities (e.g. cancer) that might put the patient at risk when following study protocols.
* No history of significant issues with known or suspected hypoglycemia or any history of "severe" hypoglycemia (requiring assistance from a third party).

Ages: 30 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katrina E Donahue, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Laura A Young, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified public use data files and documentation will allow researchers to have access to the final research data collected for this study. Care will be taken to remove indirect identifiers or other information that could result in the inadvertent disclosure of participants' identities due to the occurrence of unusual data elements. The public use database will be stored at the University of North Carolina's Sheps Center for Health Services Research. Researchers who would like access to the public-use data files for this study must enter into a data use agreement to ensure that the information will be used solely for statistical analysis or research reporting purposes. The project co-investigators in conjunction with the project manager will review requests for data and authorize provision of instructions and passwords needed to download the dataset. The public use data will be available after submission of the publication reporting the main trial findings.

REFERENCES:
- [Background] Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009 Jan;32(1):193-203. doi: 10.2337/dc08-9025. Epub 2008 Oct 22. PMID 18945920
- [Background] Quality of life in type 2 diabetic patients is affected by complications but not by intensive policies to improve blood glucose or blood pressure control (UKPDS 37). U.K. Prospective Diabetes Study Group. Diabetes Care. 1999 Jul;22(7):1125-36. doi: 10.2337/diacare.22.7.1125. PMID 10388978
- [Background] Vijan S. In the clinic. Type 2 diabetes. Ann Intern Med. 2010 Mar 2;152(5):ITC31-15; quiz ITC316. doi: 10.7326/0003-4819-152-5-201003020-01003. PMID 20194231
- [Background] American Diabetes Association. Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S14-80. doi: 10.2337/dc14-S014. No abstract available. PMID 24357209
- [Background] Towfigh A, Romanova M, Weinreb JE, Munjas B, Suttorp MJ, Zhou A, Shekelle PG. Self-monitoring of blood glucose levels in patients with type 2 diabetes mellitus not taking insulin: a meta-analysis. Am J Manag Care. 2008 Jul;14(7):468-75. PMID 18611098
- [Background] Allemann S, Houriet C, Diem P, Stettler C. Self-monitoring of blood glucose in non-insulin treated patients with type 2 diabetes: a systematic review and meta-analysis. Curr Med Res Opin. 2009 Dec;25(12):2903-13. doi: 10.1185/03007990903364665. PMID 19827909
- [Background] Farmer AJ, Perera R, Ward A, Heneghan C, Oke J, Barnett AH, Davidson MB, Guerci B, Coates V, Schwedes U, O'Malley S. Meta-analysis of individual patient data in randomised trials of self monitoring of blood glucose in people with non-insulin treated type 2 diabetes. BMJ. 2012 Feb 27;344:e486. doi: 10.1136/bmj.e486. PMID 22371867
- [Derived] Kowitt SD, Donahue KE, Fisher EB, Mitchell M, Young LA. How is neighborhood social disorganization associated with diabetes outcomes? A multilevel investigation of glycemic control and self-reported use of acute or emergency health care services. Clin Diabetes Endocrinol. 2018 Oct 19;4:19. doi: 10.1186/s40842-018-0069-0. eCollection 2018. PMID 30377539
- [Derived] Young LA, Buse JB, Weaver MA, Vu MB, Mitchell CM, Blakeney T, Grimm K, Rees J, Niblock F, Donahue KE; Monitor Trial Group. Glucose Self-monitoring in Non-Insulin-Treated Patients With Type 2 Diabetes in Primary Care Settings: A Randomized Trial. JAMA Intern Med. 2017 Jul 1;177(7):920-929. doi: 10.1001/jamainternmed.2017.1233. PMID 28600913
- [Derived] Young LA, Buse JB, Weaver MA, Vu MB, Reese A, Mitchell CM, Blakeney T, Grimm K, Rees J, Donahue KE. Three approaches to glucose monitoring in non-insulin treated diabetes: a pragmatic randomized clinical trial protocol. BMC Health Serv Res. 2017 May 25;17(1):369. doi: 10.1186/s12913-017-2202-7. PMID 28545493
- See also: National diabetes information clearinghouse — https://www.niddk.nih.gov/health-information/diabetes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified via the electronic health record (EHR) and were called to determine if they met inclusion criteria that not available from the EHR: did not plan to move or get pregnant in the next year, did not see an endocrinologist for their diabetes care, and was a patient of record in one of the 15 participating clinics.
Groups:
- No Testing: No SMBG testing
- SMBG Standard Messaging: Daily SMBG with standard messaging
- SMBG Enhanced Messaging: Daily SMBG with enhanced messaging
Period: Overall Study
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Started | 152 | 150 | 148
Completed | 147 | 142 | 139
Not Completed | 5 | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging | Total
Number analyzed (Participants) | 152 | 150 | 148 | 450
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (11.6) | 59.9 (11.4) | 60.7 (11.5) | 60.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 83 | 66 | 227
  Male | 74 | 67 | 82 | 223
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 2 | 8
  Not Hispanic or Latino | 148 | 147 | 146 | 441
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 2 | 3
  Asian | 3 | 2 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 42 | 55 | 51 | 148
  White | 104 | 89 | 86 | 279
  More than one race | 2 | 1 | 2 | 5
  Unknown or Not Reported | 0 | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 152 | 150 | 148 | 450

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in % Hemoglobin A1c From Baseline at 52 Weeks
Description: Absolute Change in Glycemic Control (% Hemoglobin A1c) from baseline at 52 weeks
Time Frame: Baseline to 52 weeks
Population: Differences in overall numbers by arm from the completed flow totals are due to the fact that not all participants were able to provide blood samples yet were able to complete all or part of the patient interview.
Measure: Mean (Standard Deviation); unit: Percent Hemoglobin A1c
Groups:
- No Testing: No Self-Monitoring of Blood Glucose (SMBG) testing
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 147 | 141 | 139
Percent Hemoglobin A1c | 0.04 (1.12) | -0.05 (1.00) | -0.10 (1.14)

2. Primary Outcome: Mean Difference in Health-related Quality of Life Scores From Baseline to 52 Weeks
Description: Change in Short Form-36 (SF-36) subscale scores (Physical and Mental subscales) from baseline to 52 weeks. The SF-36 is a widely used measure of health-related quality of life. Each subscale score ranges from 0 - 100, with 100 being the best quality of life score.
Time Frame: Baseline to 52 weeks
Population: Differences in overall numbers by arm from the completed flow totals are due to the fact that not all participants were able to complete the SF-36, yet did provide blood samples for A1c testing.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 143 | 142 | 135
Units on a scale
  SF-36: Physical Score | -.43 (6.86) | .07 (6.77) | -.35 (6.95)
  SF-36: Mental Score | -.94 (7.46) | -.71 (7.72) | -1.39 (6.85)

3. Secondary Outcome: Change in Problem Areas in Diabetes Scores From Baseline to 52 Weeks
Description: The change from baseline Problem Areas in Diabetes (PAID) scores will be assessed at 52 weeks. The PAID is a widely used tool to assess psychological and social stress associated with diabetes. The PAID scores range from 0 to 100, with 100 indicating the most distress.
Time Frame: Baseline to 52 weeks
Population: Differences in overall numbers by arm from the completed flow totals are due to the fact that not all participants were able to complete this scale, yet did provide blood samples for A1c testing and vice versa.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 143 | 142 | 135
units on a scale | -1.97 (15.44) | -4.01 (12.16) | -3.84 (13.53)

4. Secondary Outcome: Change in Diabetes Symptom Checklist- Revised (DSC-R) Overall Score From Baseline to 52 Weeks
Description: Change in diabetes-related symptom frequency and perceived severity from baseline at 52 weeks using the Diabetes Symptom Checklist-Revised. Overall score ranges from 0 to 170, with 170 indicating the worse symptom severity.
Time Frame: Baseline to 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 143 | 142 | 135
units on a scale | 2.15 (14.37) | -2.36 (15.37) | .53 (14.78)

5. Secondary Outcome: Change in Summary of Diabetes Self Care Activities (SDCA) Subscales From Baseline to 52 Weeks
Description: Change in the SDCA subscales (general diet, specific diet, exercise, blood sugar testing, and foot care), a multidimensional measure of diabetes self-management activities, from baseline at 52 weeks will be assessed. For each subscale, the score is the mean number of days specified subscale activities occurred. Each subscale ranges from 0 to 7, with 7 the best score possible.
Time Frame: Baseline to 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 143 | 142 | 135
units on a scale
  General diet | .24 (2.22) | .45 (2.26) | .17 (2.11)
  Specific diet | .11 (1.80) | -.03 (1.64) | .09 (1.70)
  Exercise | .30 (2.07) | .22 (2.10) | .37 (2.48)
  Blood sugar testing | -1.46 (2.83) | 2.94 (3.23) | 2.81 (3.30)
  Foot care | .10 (2.32) | .27 (2.44) | .39 (2.22)

6. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire Subscale Scores From Baseline to 52 Weeks
Description: Change from baseline patient satisfaction with treatment at 52 weeks using the Diabetes Treatment Satisfaction Questionnaire subscales, overall satisfaction and satisfaction with blood glucose control. For overall satisfaction, the range is 0-36, with 36 (high score) being the most satisfied. For satisfaction with blood glucose control, the subscale range is 0 to 12, with 0 (low score) indicating the most satisfaction.
Time Frame: Baseline to 52 weeks
Population: Differences in overall numbers by arm from the completed flow totals are due to the fact that not all participants were able to complete this scale, yet did provide blood samples for A1c testing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 133 | 138 | 135
units on a scale
  Overall satisfaction | -.16 (6.26) | .67 (4.95) | -.28 (5.84)
  Perceived blood glucose control | .01 (2.96) | -.12 (3.08) | -.31 (2.93)

7. Secondary Outcome: Change Diabetes Empowerment Scale - Short Form (DES-SF) From Baseline to 52 Weeks
Description: Changes in diabetes-specific self-efficacy using the Diabetes Empowerment Scale - Short Form from baseline at 52 weeks. The scale ranges from 1 to 5, with 5 indicating most empowered.
Time Frame: Baseline to 52 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 143 | 141 | 135
units on a scale | .08 (.53) | .11 (.50) | .20 (.49)

8. Secondary Outcome: Change in Patient-Provider Communication From Baseline to 52 Weeks
Description: Change from baseline patient perception of communication with their provider at 52 weeks using the Communication Assessment Tool (CAT). Scale scores range from 1 to 5, with 5 being the best communication.
Time Frame: Baseline to 52 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 141 | 142 | 134
units on a scale | .03 (.68) | -.02 (.65) | .01 (.75)

9. Secondary Outcome: Hypoglycemia Frequency
Description: Number of participants with hypoglycemia events for the 52 week intervention period.
Time Frame: Baseline to 52 weeks
Population: Differences in overall numbers by arm from the completed flow totals are due to the fact that not all participants were able to provide information for this measure, yet did provide blood samples for A1c testing and vice versa.
Measure: Count of Participants; unit: Participants
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 144 | 142 | 135
Participants | 3 | 2 | 3

10. Secondary Outcome: Baseline Health Care Utilization and at 52 Weeks
Description: Primary care visits, hospitalization, urgent care, and emergency room and emergency medical service (EMS) visits recorded at baseline and 52 weeks.
Time Frame: Baseline and 52 weeks
Population: Differences in overall numbers by arm from the completed flow totals are due to the fact that not all participants were able provide this information, yet did provide blood samples for A1c testing and vice versa.
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 144 | 142 | 135
number of events
  Primary care provider visits (baseline) | 4.0 (3.0) | 3.4 (1.6) | 3.7 (2.3)
  Primary care provider visits (follow-up)) | 3.5 (2.4) | 3.5 (2.8) | 3.5 (1.8)
  Urgent Care visits - baseline | .5 (1.3) | .4 (1.0) | .4 (.8)
  Urgent Care visits - follow-up | .3 (.7) | .3 (.8) | .3 (.6)
  Emergency room visits - baseline | .5 (1.3) | .2 (.5) | .5 (1.3)
  Emergency room visits - follow-up | .3 (.7) | .3 (.6) | .4 (1.0)
  Overnight hospitalization - baseline | .1 (.3) | .1 (.4) | .1 (.3)
  Overnight hospitalization - follow-up | .1 (.3) | .1 (.4) | .1 (.4)
  EMS called - baseline | .2 (.6) | .1 (.2) | .1 (.2)
  EMS called - follow-up | .1 (.3) | 0.0 (.2) | .1 (.3)

11. Secondary Outcome: Number of Participants on Specified Diabetes Medications at Baseline and Follow-up
Description: Number of participants taking each of the following medications at baseline and follow-up: metformin, sulfonylurea, glinides, Glucagon-like peptide-1 (GLP-1), Thiazolidinediones (TZD), and dipeptidyl peptidase IV (DPP-IV).
Time Frame: Baseline and 52 weeks
Population: Medication regimens vary among patients.
Measure: Count of Participants; unit: Participants
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Number analyzed (Participants) | 152 | 150 | 148
Participants
  Metformin - baseline | 123 | 115 | 120
  Metformin - follow-up: number analyzed (Participants) | 148 | 150 | 148
  Metformin - follow-up | 124 | 114 | 111
  Sulfonylurea - baseline | 50 | 49 | 60
  Sulfonylurea - follow-up | 56 | 63 | 65
  Glinides - baseline | 1 | 1 | 0
  Glinides - follow-up | 0 | 1 | 0
  GLP-1 - baseline | 5 | 2 | 10
  GLP-1 - follow-up | 6 | 6 | 11
  TZD - baseline | 8 | 3 | 10
  TZD - follow-up | 7 | 1 | 14
  DPP-IV - baseline | 12 | 11 | 17
  DPP-IV - follow-up | 16 | 14 | 17

ADVERSE EVENTS:
Time Frame: From Randomization date until Final Visit date: 52 weeks +-6 weeks
Arm/Group | No Testing | SMBG Standard Messaging | SMBG Enhanced Messaging
Serious Adverse Events (participants affected / at risk) | 2/152 | 0/150 | 1/148
Other Adverse Events (participants affected / at risk) | 6/152 | 9/150 | 10/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Testing (N=152) | SMBG Standard Messaging (N=150) | SMBG Enhanced Messaging (N=148)
Death (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Death (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Severe Hypoglycemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Testing (N=152) | SMBG Standard Messaging (N=150) | SMBG Enhanced Messaging (N=148)
Hospitalization (General disorders) | 6 (6) | 9 (9) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No